CLINICAL TRIAL: NCT01156493
Title: Randomized Trial of Hydrolyzed Protein Premature Formula
Brief Title: Hydrolized Protein Formula for Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Teresa del Moral, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20090579
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2015-11

CONDITIONS: Prematurity
Keywords: feeding intolerance; prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Protein Hydrolized Formula
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Standard Formula
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protein Hydrolyzed Formula (Experimental): Infants assigned to this group will receive HP formula when breast milk not available or indicated to receive formula by the attending physician
  Interventions: Other: Protein Hydrolyzed Premature Formula
- Control (No Intervention): Infants in this group will receive standard prematrue formula when no breast milk available or indicated by the attending physician

INTERVENTIONS:
Other: Protein Hydrolyzed Premature Formula — Infants will be fed with a protein hydrolyzed premature formula until they reach full feeds
  Arms: Protein Hydrolyzed Formula

SUMMARY:
Premature infants fed with a protein hydrolyzed formula will have better tolerance needing shorter time to achieve full feeds when compared to those fed with an intact protein formula.

DETAILED DESCRIPTION:
The study formula is a 100% whey protein partially hydrolyzed (vs 60/40 Whey:Casein ratio of regular premature formulas) Because the tolerance and availability of breast milk is not predictable at the time of enrollment all the eligible premature infants will be randomized and assigned to the study or control group. Infants will receive formula, either because breast milk is not available or because indicated by the attending physician and switched to formula, They will be fed, depending of the group to what they are assigned, with either the PH formula for the study group or regular premature formula for the control group.

Randomization and blinding All eligible infants with parental consent will be randomized to either the study group to receive protein hydrolyzed formula (PH group) or to the control group to receive standard premature formula. Randomization will be stratified by 2 birth weight categories (500-1000 g and 1001-1500 g). The purpose of such stratification is to avoid imbalance between groups for factors that may influence outcome and is based on the different morbidity in different birth weight categories.

Masked randomization will be performed in a way that avoids the possibility of knowledge of treatment assignment at the time that eligibility is assessed and consent is sought. Only the person in charge of preparing the control or study formula will be aware of the infant's assignment group. Caregivers will remain masked to treatment group.

Study population Preterm newborns admitted to the neonatal intensive care unit with a birth weight 500-1500 g and who survive more than 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight between 500 -1500g and < 32 weeks GA who survive more than 3 days.
* Has not yet started enteral full feeds.
* Study explained and parent/caregiver demonstrating understanding of the given information.
* Informed consent signed.

Exclusion Criteria:

* Chromosomal anomalies.
* Major congenital anomalies (complex cardiac anomalies, congenital hydrocephalus, renal dysplasia).
* Congenital (e.g. jejunal atresia) and acquired (e.g. GI perforation) gastrointestinal pathology precluding oral feed and/or requiring major surgical or medical intervention.
* Parental refusal.
* Prior enrollment into a conflicting clinical trial. Conflicting clinical trial will be those in which the intervention could modify the outcome of the present study, for example studies aimed to accelerate feeds and or improve tolerance.

Ages: 3 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Time to achieve full feeds | Average 1 to 3 weeks of life
  Number of days from initiating oral feeds to achieve full feeds

SECONDARY OUTCOMES:
Postnatal days to achieve full feeds | Average: 1- 3 weeks of age
  number of days from birth to achieve full feeds

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Del Moral, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami/Holtz Children's Hospital/Neonatal Intensive Care Unit, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No